CLINICAL TRIAL: NCT06822153
Title: A Single-center, Randomized, Open-label, Placebo-controlled Phase I Clinical Trial Was Conducted to Evaluate the Pharmacokinetics and QT Interval Effects of a Single Intravenous Injection of Methoxyethyl Etomidate Hydrochloride in Healthy Subjects
Brief Title: Clinical Trial of the Effect of Methoxyethyl Etomidate Hydrochloride on the QT Interval of the Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET-26-HCL-CP-002
Record Dates: First submitted 2025-01-24; First posted 2025-02-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: QT Interval, Variation in
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose group (Other): Placebo+ET-26 0.8mg/kg
  Interventions: Drug: ET-26 0.8mg/kg(low-dose) group
- High dose group (Other): Placebo+ET-26 2.8mg/kg
  Interventions: Drug: ET-26 2.8mg/kg(high dose) group

INTERVENTIONS:
Drug: ET-26 0.8mg/kg(low-dose) group — In a 2:1 ratio, Placebo was administered with normal saline and ET-26 0.8mg/kg for a duration of 60 ±5 seconds.
  Arms: low-dose group
Drug: ET-26 2.8mg/kg(high dose) group — In a 2:1 ratio, Placebo was administered with normal saline and ET-26 2.8mg/kg for a duration of 60 ±5 seconds.
  Arms: High dose group

SUMMARY:
A single intravenous injection of 0.8mg/kg or 2.8mg/kg Et-26-hcl was given to 18 subjects. The effect of plasma concentration on QT interval was evaluated by C-QTc effect model, and the pharmacokinetic characteristics and safety of ET-26 and etomidate acid were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female subjects;
2. Age: 18-45 years old;
3. Body weight: body mass index (BMI) between 19.0 and 28.0 kg/m2, with a body weight of at least 50 kg for male subjects and 45 kg for female subjects;
4. voluntarily sign informed consent;
5. Subjects were able to communicate well with investigators and complete the trial in accordance with the protocol.

Exclusion Criteria:

-

Auxiliary examination:

1. those with clinically significant abnormalities in comprehensive physical examination, vital signs, and laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, serum cortisol);
2. potentially difficult airway (modified Mallampati score III-IV);
3. abnormal and clinically significant hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia, or hypocalcemia as judged by the investigator;
4. clinically significant abnormal 12-lead ECG, QTcF≥450 ms, PR interval ≥200 ms, QRS complex duration ≥120ms;
5. hepatitis B surface antigen, hepatitis C antibody, HIV antibody or syphilis antibody positive;

   Medication history:
6. use of any drugs that inhibit or induce hepatic drug-metabolizing enzymes within 30 days before screening (see Appendix 1 for details);
7. Use of any known QT-prolonging medication within 30 days before screening (see Appendix 1 for details);
8. use of any prescribed medication within 14 days before dose;
9. use of over-the-counter medications, Chinese herbal medicines, or food supplements such as vitamins and calcium supplements within 7 days before administration;

   History of disease and surgery:
10. have a history of any clinically serious diseases or diseases or conditions considered by the investigators to be likely to affect the results of the trial, including but not limited to a history of circulatory, respiratory, endocrine, nervous, digestive, urinary, or hematologic, immune, psychiatric, or metabolic diseases;
11. with a history of adrenal insufficiency, adrenal tumors, or hereditary heme biosynthesis disorders;
12. a history of severe cardiovascular disease, including but not limited to organic heart disease, such as heart failure, myocardial infarction, angina pectoris, or malignant arrhythmia, as judged by the investigator; Such as a history of torssion ventricular tachycardia, ventricular tachycardia, long QT syndrome or symptoms of long QT syndrome and family history (as indicated by genetic evidence or sudden death of a close relative at a young age due to cardiac causes);
13. underwent any surgery within 6 months before screening;
14. allergic constitution, such as known allergic history to two or more substances; Or who, as judged by the investigator, may be allergic to the trial drug or its excipients;

    Living habits:
15. heavy drinking or regular drinking in the 6 months before screening, i.e. drinking more than 14 units of alcohol per week (1 unit =360 mL of beer or 45 mL of 40% spirits or 150 mL of wine); Or with a positive alcohol breath test during the screening period;
16. used nicotine-containing products between 3 months before screening and study enrollment;
17. with drug abuse or drug abuse history within 3 months before screening; Or the urine drug test was positive in the screening period;
18. habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages and inability to quit during the trial;

    Others:
19. who had difficulty in blood collection or could not tolerate blood collection by venipuncture;
20. participated in any other clinical trial (including drug and device clinical trials) within 3 months before screening;
21. vaccinated within 1 month before screening or planned to be vaccinated during the trial period;
22. pregnant or lactating women;
23. during the trial and within half a year after the completion of the trial, or those who do not agree that the subjects and their spouses should take strict contraceptive measures during the trial and within half a year after the completion of the trial (see Appendix 4 for details);
24. had blood loss or donation > 400 mL within 3 months before screening, or received blood transfusion within 1 month;
25. had any factors considered by the investigator to preclude participation in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | from 1 hour before administration of et-26 until 24 hours after the end of administration.
  Cmax

SECONDARY OUTCOMES:
MOAA/S | up to 10 minutes after drug administration
  modified observer's assessment of alert（MOAA/S） score: The lowest score was 0, indicating full anesthetic sedation, and the highest score was 5, indicating full consciousness.
Eyelash reflex | up to 2 minutes after drug administration
  Gently touching the subject's eyelashes with a cotton swab can cause the subject to blink, that is, there is an eyelash reflex. When the eyelash reflex disappears, the patient has entered a state of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wen, Master, Principal Investigator — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China